CLINICAL TRIAL: NCT04624607
Title: Transspinal-Transcortical Paired Stimulation for Neuroplasticity and Recovery After SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: College of Staten Island, the City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-0261; C32095GG (Other Grant/Funding Number: New York State Department of Health Spinal Cord Injury Research Board)
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Spinal Cord Injuries; Paraplegia, Spinal; Tetraplegia/Tetraparesis
Keywords: Spinal Cord Injury; Locomotor Training; Neuromodulation; Paired-Associative Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Intervention Model Description: Individuals with Spinal Cord Injury will be assigned to receive robotic gait training with the Lokomat combined with paired non-invasive thoracolumbar transspinal stimulation and non-invasive brain stimulation.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transspinal-transcortical paired-associative stimiulation combined with robotic gait training (Experimental): Robotic gait training will be administered along with paired non-invasive transspinal stimulation over the thoracolumbar region and non-invasive brain stimulation during assisted stepping.
  Interventions: Device: Transspinal-transcortical paired-associative stimiulation combined with robotic gait training
- Transcortical-transspinal paired-associative stimiulation combined with robotic gait training (Experimental): Robotic gait training will be administered along with paired non-invasive brain stimulation and non-invasive transspinal stimulation over the thoracolumbar region during assisted stepping.
  Interventions: Device: Transcortical-transspinal paired-associative stimiulation combined with robotic gait training

INTERVENTIONS:
Device: Transspinal-transcortical paired-associative stimiulation combined with robotic gait training — Individuals with spinal cord injury will receive 20 daily sessions of robotic gait training. During assisted stepping, they will receive also paired non-invasive transspinal stimulation and non-invasive brain stimulation during the stance phase of gait. Before and after training standardized clinical and neurophysiological tests will be used to assess recovery of sensorimotor function.
  Arms: Transspinal-transcortical paired-associative stimiulation combined with robotic gait training
Device: Transcortical-transspinal paired-associative stimiulation combined with robotic gait training — Individuals with spinal cord injury will receive 20 daily sessions of robotic gait training. During assisted stepping, they will receive also paired non-invasive brain stimulation and non-invasive transspinal stimulation during the stance phase of gait. Before and after training standardized clinical and neurophysiological tests will be used to assess recovery of sensorimotor function.
  Arms: Transcortical-transspinal paired-associative stimiulation combined with robotic gait training

SUMMARY:
People with spinal cord injury (SCI) have motor dysfunction that results in substantial social, personal, and economic costs. Uncontrolled muscle spasticity and motor dysfunction result in disabilities that significantly reduce quality of life. Several rehabilitation interventions are utilized to treat muscle spasticity and motor dysfunction after SCI in humans. However, because most interventions rely on sensory afferent feedback that is interpreted by malfunctioned neuronal networks, rehabilitation efforts are greatly compromised. On the other hand, changes in the function of nerve cells connecting the brain and spinal cord have been reported following repetitive electromagnetic stimulation delivered over the head and legs or arms at specific time intervals. In addition, evidence suggests that electrical signals delivered to the spinal cord can regenerate spinal motor neurons in injured animals. A fundamental knowledge gap still exists on neuroplasticity and recovery of leg motor function in people with SCI after repetitive transspinal cord and transcortical stimulation. In this project, it is proposed that repetitive pairing of transspinal cord stimulation with transcortical stimulation strengthens the connections between the brain and spinal cord, decreases ankle spasticity, and improves leg movement. People with motor incomplete SCI will receive transspinal - transcortical paired associative stimulation at rest and during assisted stepping. The effects of this novel neuromodulation paradigm will be established via clinical tests and noninvasive neurophysiological methods that assess the pathways connecting the brain with the spinal cord.

DETAILED DESCRIPTION:
Motor dysfunction after SCI results in substantial personal, social, and economic costs. Secondary complications related to muscle spasticity and motor dysfunction significantly reduce quality of life. Rehabilitation efforts are compromised because most therapeutic interventions rely heavily on sensory afferent feedback that is interpreted by malfunctioned neuronal networks. On the other hand, electrical signals delivered over the spine regenerate neurons of the spinal cord in injured animals, and paired associative stimulation produces enduring neuronal plasticity in healthy and injured humans and animals. A fundamental knowledge gap still exists on induction of functional neuroplasticity and recovery of leg motor function following repetitive pairing of transspinal cord stimulation with transcortical stimulation in people with motor incomplete SCI. Our central working hypothesis is that transspinal cord stimulation paired with transcortical stimulation strengthens corticospinal neuronal connections, decreases ankle spasticity, and improves leg motor function. This notion is based on the concept tested in the applicant's laboratory that this novel stimulation paradigm potentiates synaptic actions and activity of spared but compromised axons providing the necessary environment for functional neuroplasticity. The rationale of this research study is that neuromodulation methods that can modify effectively the input-output relations of cortical and spinal neuronal pathways in people with motor incomplete SCI are needed. Based on strong preliminary data, two specific aims will be addressed: Specific Aim 1: Establish induction of transspinal-transcortical paired associative stimulation (PAS) neuroplasticity and improvements in leg sensorimotor function in people with motor incomplete SCI when PAS is administered during robotic-assisted gait training. Cortical and corticospinal neuronal circuits via state-of-the-art neurophysiological methods in seated (Aim 1A), soleus H-reflex excitability during assisted stepping (Aim 1B), and sensorimotor function evaluated via standardized clinical tests (Aim 1C) will be assessed before and after 15 sessions of transspinal-transcortical PAS delivered with subjects supine. Specific Aim 2: Establish induction of transcortical-transspinal PAS neuroplasticity and improvements in leg sensorimotor function in people with motor incomplete SCI when PAS is administered during assisted stepping. Cortical and corticospinal neuroplasticity via state-of-the-art neurophysiological methods in seated (Aim 2A), soleus H-reflex excitability during assisted stepping (Aim 2B), and leg sensorimotor function evaluated via standardized clinical tests (Aim 2C) will be assessed before and after 15 sessions of transspinal-transcortical PAS delivered during assisted stepping. It is hypothesized that transspinal-transcortical PAS delivered at rest or during assisted stepping strengthens corticospinal connections, increases spinal inhibition, decreases ankle spasticity, and improves leg motor function. Further, transspinal-transcortical PAS delivered during assisted stepping normalizes the abnormal phase-dependent soleus H-reflex modulation commonly observed during stepping in people with motor incomplete SCI. To test the project hypotheses, 12 people with motor incomplete SCI will receive 20 sessions of transspinal-transcortical or transcortical-transspinal PAS during assisted stepping. In people with SCI, and assess improvements in leg motor function with standardized clinical tests. In all subjects, assessments of neuroplasticity in cortical, corticospinal, and spinal neuronal networks will be administered. These results will advance considerably the field of spinal cord research and change the standard of care because there is great potential for development of novel and effective rehabilitation strategies to manage spasticity and improve motor function after SCI in humans.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of motor incomplete spinal cord injury (SCI).
* SCI is above thoracic 12 vertebra.
* Absent permanent ankle joint contractures.
* SCI occurred 6 months before enrollment to the study.

Exclusion Criteria:

* Supraspinal lesions
* Neuropathies of the peripheral nervous system
* Degenerative neurological disorders
* Presence of pressure sores
* Urinary tract infection
* Neoplastic or vascular disorders of the spine or spinal cord
* Pregnant women or women who suspect they may be or may become pregnant
* People with cochlear implants, pacemaker, and implanted simulators
* People with history of seizures
* People with implanted Baclofen pump

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Plasticity of cortical and corticospinal neural circuits | 3 years
  Neurophysiological tests probing cortical and corticospinal excitability will be measured before and after the intervention. Single-pulse transcranial magnetic stimulation (TMS) will be used to assemble the recruitment curve of motor evoked potentials, and paired-pulse TMS will be used to probe changes in cortical inhibitory and facilitatory neuronal circuits.
Plasticity of spinal neural cicuits | 3 years
  Neurophysiological tests probing spinal reflex excitability will be measured before and after each intervention by posterior tibial and sural nerves stimulation during Lokomat-assisted stepping depicting the amplitude modulation of the soleus H-reflex, tibialis anterior flexor reflex, and interlimb reflexes.

SECONDARY OUTCOMES:
Sensorimotor leg motor function | 3 years
  Manual muscle test and leg sensation based on American Spinal Injury Association
Walking function | 3 years
  Two-minute walk test and 10 meter timed test

CONTACTS AND LOCATIONS:
Overall Officials: Maria Knikou, PT, PhD, Principal Investigator — College of Staten Island, City University of New York
Locations (1):
- Department of Physical Therapy, College of Staten Island, City University of New York, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dixon L, Ibrahim MM, Santora D, Knikou M. Paired associative transspinal and transcortical stimulation produces plasticity in human cortical and spinal neuronal circuits. J Neurophysiol. 2016 Aug 1;116(2):904-16. doi: 10.1152/jn.00259.2016. Epub 2016 Jun 8. PMID 27281748
- [Background] Knikou M. Spinal Excitability Changes after Transspinal and Transcortical Paired Associative Stimulation in Humans. Neural Plast. 2017;2017:6751810. doi: 10.1155/2017/6751810. Epub 2017 Oct 16. PMID 29123926
- [Background] Knikou M. Functional reorganization of soleus H-reflex modulation during stepping after robotic-assisted step training in people with complete and incomplete spinal cord injury. Exp Brain Res. 2013 Jul;228(3):279-96. doi: 10.1007/s00221-013-3560-y. Epub 2013 May 25. PMID 23708757
- [Background] Stefan K, Kunesch E, Cohen LG, Benecke R, Classen J. Induction of plasticity in the human motor cortex by paired associative stimulation. Brain. 2000 Mar;123 Pt 3:572-84. doi: 10.1093/brain/123.3.572. PMID 10686179
- [Background] Smith AC, Mummidisetty CK, Rymer WZ, Knikou M. Locomotor training alters the behavior of flexor reflexes during walking in human spinal cord injury. J Neurophysiol. 2014 Nov 1;112(9):2164-75. doi: 10.1152/jn.00308.2014. Epub 2014 Aug 13. PMID 25122715
- [Background] Field-Fote EC, Roach KE. Influence of a locomotor training approach on walking speed and distance in people with chronic spinal cord injury: a randomized clinical trial. Phys Ther. 2011 Jan;91(1):48-60. doi: 10.2522/ptj.20090359. Epub 2010 Nov 4. PMID 21051593
- [Background] Smith AC, Rymer WZ, Knikou M. Locomotor training modifies soleus monosynaptic motoneuron responses in human spinal cord injury. Exp Brain Res. 2015 Jan;233(1):89-103. doi: 10.1007/s00221-014-4094-7. Epub 2014 Sep 10. PMID 25205562
- [Background] Taylor JL, Martin PG. Voluntary motor output is altered by spike-timing-dependent changes in the human corticospinal pathway. J Neurosci. 2009 Sep 16;29(37):11708-16. doi: 10.1523/JNEUROSCI.2217-09.2009. PMID 19759317
- [Background] Song S, Miller KD, Abbott LF. Competitive Hebbian learning through spike-timing-dependent synaptic plasticity. Nat Neurosci. 2000 Sep;3(9):919-26. doi: 10.1038/78829. PMID 10966623
- [Background] Thomas SL, Gorassini MA. Increases in corticospinal tract function by treadmill training after incomplete spinal cord injury. J Neurophysiol. 2005 Oct;94(4):2844-55. doi: 10.1152/jn.00532.2005. Epub 2005 Jul 6. PMID 16000519
- [Derived] Pulverenti TS, Zaaya M, Knikou M. Brain and spinal cord paired stimulation coupled with locomotor training affects polysynaptic flexion reflex circuits in human spinal cord injury. Exp Brain Res. 2022 Jun;240(6):1687-1699. doi: 10.1007/s00221-022-06375-x. Epub 2022 May 6. PMID 35513720